CLINICAL TRIAL: NCT06236763
Title: Comparison of the TOFscan Simultaneous Measures at the Thumb and the First Toe During Recovery of Neuromuscular Function Following Rocuronium Administration
Brief Title: Comparison of Neuromuscular Recovery at the Hand and Foot
Status: Recruiting | Type: Observational
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Louis Philippe Fortier, MD, MSc, Associate Professor, Anesthesiologist, Chief officer perioperative and surgical activities, Department of Anesthesiology and Pain Medicine at University of Montréal, Ciusss de L'Est de l'Île de Montréal
Other Study IDs: 2024-3609
Record Dates: First submitted 2024-01-16; First posted 2024-02-01 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation and control: Two accelerometers will be applied on each patient; observation (foot) and control (hand, also the gold standard). Agreement values will be compared between these two monitors.
  Interventions: Device: TOFscan foot

INTERVENTIONS:
Device: TOFscan foot — TOFscan will be applied on the foot and recovery from neuromuscular blockade will be observed over time. These will be compared with the control (TOFscan at the hand) on the same patient (gold standard monitor).

SUMMARY:
Gold standard for neuromuscular blockade evaluation is accelerometry in three dimensions at the thumb. There are many times that measurement at the hand can be falsely under-estimated intraoperatively secondary to constriction of the upper extremities. We believe that installing the same accelerometer at the first toe will give us similar readings for both neuromuscular blockade and recovery from rocuronium administration. This study focuses on agreement values between two accelerometers installed on the hand and at on the foot.

DETAILED DESCRIPTION:
The development of advanced competence in laparoscopic surgery, robotic surgery and the broadening of indications for partial or total laparoscopy techniques created a novel environment where patients need to be deeply paralyzed and positioned in form fitting mattresses to ensure high quality exposure and security in extreme positioning. It is now undisputed that clinical evaluation done any other way than by a objective neuromuscular function monitor may produce faulty conclusions. The elements of the operating setup force anesthesiologists to adapt the way they monitor muscle relaxation since the hands are generally not available for neuromuscular function monitoring. In order to measure properly the level of residual paralysis, the thumb must be able to move freely in a device creating a light preloading on the adductor pollicis allowing to evaluate the force generated during standardized stimulation through accelerometry, the TOFscan device. The corrugator supercilli and orbicularis oculi muscles, an alternate positioning for the accelerometer is sometimes the fallback spot for monitoring. The problem with that muscle is that it does not have the same time curve sensitivity to muscle relaxant than the perilaryngeal muscle have. The investigators are looking for a good representation of the level of patency of the perilaryngeal muscle to ensure that the patient will be able to breath normally after extubation, they must turn to another target. Previous observations have suggested that the monitoring of the hallux flexor muscle could represent a valid alternative. The confirmation of this hypothesis would allow for easy, reproducible, evaluation of the level of muscle relaxation at the perilaryngeal muscles, helping to procure safer conditions for tracheal extubation. Neuromuscular blocking agents (NMBAs) are administered by anesthesiologists during general anesthesia to facilitate endotracheal intubation and/or surgical conditions. Postoperative residual neuromuscular blockade (rNMB), is an adverse event frequently observed after extubation in the postanesthesia care unit (PACU) after surgery. rNMB is associated with upper airway obstruction, reduced pharyngeal muscle coordination, decreased functional residual capacity, and impaired hypoxic ventilatory response and may lead to critical cardiopulmonary complications. To prevent those complications, monitoring NMBAs activity and timely and adequate dosage of reversal agents necessitate precise and valid monitoring.

The current literature supports the exclusive use of quantitative measurements of residual paralysis, subjective monitoring caries to much error in evaluating the level of blockade and is responsible for PACU residual paralysis and its complications. It is well accepted that no amount of rNMB is acceptable (TOF < 1) around extubation periods, a necessary step to ensure safety that relies on timely and correct dosage of the reversal agents.

When TOFscan measures are done on partially mobile thumbs, or transducers positioned in non-optimal fashion, the measure observed (deep blockade) will either delay the reversal procedure because of presumed very deep level paralysis or suggest high doses of reversal agents at a significant cost.

The investigators are confident that validating the measures done at the hallux flexor will allow for easy, relevant and valid estimation of residual paralysis and create a safer environment for muscle relaxation reversal and extubation.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3 patients
* Elective surgery
* Undergoing general anesthesia with rocuronium induced NMB
* BMI < 36 kg.m-2
* Age > 18 years old
* French or English speaking patient

Exclusion Criteria:

* Renal or hepatic dysfunction
* Obstructive sleep apnea requiring continuous positive airway pressure (CPAP) machine
* Neuromuscular disease
* Peripheral arterial disease (suspected, known or investigated)
* Calcium channel anomalies
* Hypothermia (< 35C)
* Hyper/hypomagnasemia
* Allergy to any drug used in the study protocol
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any patient scheduled for more than 2 hours extra cavitary surgery where muscle relaxation spontaneous reversal will not interfere with the completion of the planned surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Time of neuromuscular blockade (NMB) recovery | 60 minutes
  Time required for train-of-four (TOF) > 0.9 for the two TOFscans

SECONDARY OUTCOMES:
Neuromuscular blockade onset | 3 minutes
  Time to train-of-four (TOF) count of 0 for both monitors
Reversal | 60 minutes
  Train-of-four ratio (TOF) immediately before reversal agent administration on both monitors
Extubation | 1 minute
  Train-of-four (TOF) ratio at extubation

CONTACTS AND LOCATIONS:
Overall Officials: 514-252-3426 Fortier, MD, Principal Investigator — Maisonneuve-Rosemont Hospital - CIUSSS de l'Est de l'Ile de Montréal
Locations (1):
- Maisonneuve-Rosemont Hospital - CIUSSS de l'Est de l'Ile de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Naguib M, Brull SJ, Johnson KB. Conceptual and technical insights into the basis of neuromuscular monitoring. Anaesthesia. 2017 Jan;72 Suppl 1:16-37. doi: 10.1111/anae.13738. PMID 28044330
- [Result] Unterbuchner C, Ehehalt K, Graf B. [Algorithm-based preventive strategies for avoidance of residual neuromuscular blocks]. Anaesthesist. 2019 Nov;68(11):744-754. doi: 10.1007/s00101-019-00677-6. German. PMID 31650189
- [Result] D'Honneur G, Guignard B, Slavov V, Ruggier R, Duvaldestin P. Comparison of the neuromuscular blocking effect of atracurium and vecuronium on the adductor pollicis and the geniohyoid muscle in humans. Anesthesiology. 1995 Mar;82(3):649-54. doi: 10.1097/00000542-199503000-00006. PMID 7879933
- [Result] Fortier LP, McKeen D, Turner K, de Medicis E, Warriner B, Jones PM, Chaput A, Pouliot JF, Galarneau A. The RECITE Study: A Canadian Prospective, Multicenter Study of the Incidence and Severity of Residual Neuromuscular Blockade. Anesth Analg. 2015 Aug;121(2):366-72. doi: 10.1213/ANE.0000000000000757. PMID 25902322
- [Result] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS. Residual neuromuscular blockade and critical respiratory events in the postanesthesia care unit. Anesth Analg. 2008 Jul;107(1):130-7. doi: 10.1213/ane.0b013e31816d1268. PMID 18635478
- [Result] Errando CL, Garutti I, Mazzinari G, Diaz-Cambronero O, Bebawy JF; Grupo Espanol De Estudio Del Bloqueo Neuromuscular. Residual neuromuscular blockade in the postanesthesia care unit: observational cross-sectional study of a multicenter cohort. Minerva Anestesiol. 2016 Dec;82(12):1267-1277. Epub 2016 May 27. PMID 27232277
- [Result] Saager L, Maiese EM, Bash LD, Meyer TA, Minkowitz H, Groudine S, Philip BK, Tanaka P, Gan TJ, Rodriguez-Blanco Y, Soto R, Heisel O. Incidence, risk factors, and consequences of residual neuromuscular block in the United States: The prospective, observational, multicenter RECITE-US study. J Clin Anesth. 2019 Aug;55:33-41. doi: 10.1016/j.jclinane.2018.12.042. Epub 2018 Dec 27. PMID 30594097
- [Result] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Shear TD, Deshur M, Benson J, Newmark RL, Maher CE. Comparison of the TOFscan and the TOF-Watch SX during Recovery of Neuromuscular Function. Anesthesiology. 2018 Nov;129(5):880-888. doi: 10.1097/ALN.0000000000002400. PMID 30130260
- [Result] Viby-Mogensen J, Jensen NH, Engbaek J, Ording H, Skovgaard LT, Chraemmer-Jorgensen B. Tactile and visual evaluation of the response to train-of-four nerve stimulation. Anesthesiology. 1985 Oct;63(4):440-3. doi: 10.1097/00000542-198510000-00015. No abstract available. PMID 4037404
- [Result] Brull SJ, Silverman DG. Visual and tactile assessment of neuromuscular fade. Anesth Analg. 1993 Aug;77(2):352-5. doi: 10.1213/00000539-199308000-00024. PMID 8394051
- [Result] Naguib M, Brull SJ, Kopman AF, Hunter JM, Fulesdi B, Arkes HR, Elstein A, Todd MM, Johnson KB. Consensus Statement on Perioperative Use of Neuromuscular Monitoring. Anesth Analg. 2018 Jul;127(1):71-80. doi: 10.1213/ANE.0000000000002670. PMID 29200077
- [Result] Kirov K, Motamed C, Dhonneur G. Differential sensitivity of abdominal muscles and the diaphragm to mivacurium: an electromyographic study. Anesthesiology. 2001 Dec;95(6):1323-8. doi: 10.1097/00000542-200112000-00008. PMID 11748387
- [Result] Plaud B, Debaene B, Donati F. The corrugator supercilii, not the orbicularis oculi, reflects rocuronium neuromuscular blockade at the laryngeal adductor muscles. Anesthesiology. 2001 Jul;95(1):96-101. doi: 10.1097/00000542-200107000-00019. PMID 11465590
- [Result] Dhonneur G, Kirov K, Slavov V, Duvaldestin P. Effects of an intubating dose of succinylcholine and rocuronium on the larynx and diaphragm: an electromyographic study in humans. Anesthesiology. 1999 Apr;90(4):951-5. doi: 10.1097/00000542-199904000-00004. PMID 10201662